CLINICAL TRIAL: NCT05406609
Title: Cost Comparison Between General Anesthesia and Regional Anesthesia in Shoulder Operations
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, dilan akyurt, Specialist of Anaesthesiology and Reanimasion, Samsun University
Other Study IDs: B.30.2.ODM.0.20.08/229-265
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Anesthesia
Keywords: cost; Regional anesthesia; Shoulder
MeSH Terms: interventions — Costs and Cost Analysis; Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- General: Shoulder surgery under general anesthesia
  Interventions: Other: Cost; Other: Time
- Regional: Shoulder surgery under regional anesthesia
  Interventions: Other: Cost; Other: Time

INTERVENTIONS:
Other: Cost — Costs of operating room, drugs and equipments which are used by anesthesia
Other: Time — Time of using operating room

SUMMARY:
Shoulder surgery can be done not only arthroscopy but also open technic. General or regional anaesthesia can be used at this surgery. Anaesthetic choice can be changed by comorbidity factors, patients or surgeons choice etc. At this study we aimed compare the general and regional anesthesia costs during operating room.

DETAILED DESCRIPTION:
General anesthesia or ultrasound guided brachial plexus blocks (interscalene, superior trunk) can be used during shoulder surgery, as our routine. In this retrospective study, the data of patients who underwent shoulder surgery under regional or general anesthesia between 01 August 2021 and 31 March 2022 (8 months) in the operating room of the Samsun University Education and Research Hospital will be investigated. The characteristics of the patients such as age, presence of additional disease, operation indication, duration of stay in the operating room, and intraoperative medical agents will be recorded. Fees for materials used for general anesthesia and regional anesthesia will be determined. A fixed cost will be determined for the use of the operating room, including the salaries of healthcare workers. After calculating the group costs between both groups, statistical analyzes will be made.

ELIGIBILITY:
Inclusion Criteria:

* Open shoulder surgery, ASA I, II and III

Exclusion CriteriaS

* shoulder Arthroscopy , used regional anesthesia for only analgesia, American society of Anesthesiologists (ASA) score IV patients, emergency

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Shoulder surgery with general anesthesia or regional anesthesia in our hospital between ASA I-II and III group patients will be included in the study
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Cost of regional and general anesthesia | 6 months
  Calculation of peroperative cost of patients undergoing shoulder surgery under general or regional anesthesia, excluding surgical materials

SECONDARY OUTCOMES:
Time | 6 months
  Measuring the time of using operating room for shoulder surgery under general or regional anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Tulgar, Study Director — Samsun University
Locations (1):
- Dilan Akyurt, Samsun, Turkey (Türkiye)

REFERENCES:
- [Background] Gonano C, Kettner SC, Ernstbrunner M, Schebesta K, Chiari A, Marhofer P. Comparison of economical aspects of interscalene brachial plexus blockade and general anaesthesia for arthroscopic shoulder surgery. Br J Anaesth. 2009 Sep;103(3):428-33. doi: 10.1093/bja/aep173. Epub 2009 Jul 8. PMID 19586958
- [Result] Hewson DW, Oldman M, Bedforth NM. Regional anaesthesia for shoulder surgery. BJA Educ. 2019 Apr;19(4):98-104. doi: 10.1016/j.bjae.2018.12.004. Epub 2019 Feb 6. No abstract available. PMID 33456877
- [Result] Komann M, Avian A, Dreiling J, Gerbershagen H, Volk T, Weinmann C, Meissner W. Association of Perioperative Regional Analgesia with Postoperative Patient-Reported Pain Outcomes and Opioid Requirements: Comparing 22 Different Surgical Groups in 23,911 Patients from the QUIPS Registry. J Clin Med. 2021 May 19;10(10):2194. doi: 10.3390/jcm10102194. PMID 34069496
- See also: Tapar H, Suren M, Kaya Z, Arıcı S, Karaman S, Kahveci M. Üst Ekstremite Periferik Blok Anestezisi Ve Komplikasyonları — https://dergipark.org.tr/en/download/article-file/81877